CLINICAL TRIAL: NCT06421168
Title: The Impact of Body Mass Index on Lung Function in Bariatric Surgery Candidates
Brief Title: Lung Function in Bariatric Surgery Candidates
Status: Completed | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Yuntao Nie, Principal Investigator, China-Japan Friendship Hospital
Other Study IDs: CJBariatric006
Record Dates: First submitted 2024-05-13; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Lung Function Decreased; Obesity
MeSH Terms: conditions — Respiratory Insufficiency; Obesity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to retrospectively investigate the impact of body mass index on lung function metrics, e.g. FEV1%, FVC%, FEV1/FVC%.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with obesity (BMI ≥ 27.5 kg/m2 according to Chinese guidelines, guidelines from the American Society for Metabolic and Bariatric Surgery and International Federation for the Surgery of Obesity and Metabolic Disorders);
* Age > 16 years;
* Complete preoperative pulmonary function tests

Exclusion Criteria:

* Patients with a history of lung surgery and/or respiratory diseases (e.g. asthma, pulmonary emphysema, and interstitial pulmonary fibrosis).

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Bariatric surgery candidates who completed lung function tests preoperatively were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1834 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
FEV1, FVC, FEV1/FVC% in class 1, 2, and 3 obesity | At the time of pulmonary function testing
  Class 1 obesity: 27.5 kg/m2 < body mass index < 32.5 kg/m2; Class 2 obesity: 32.5 kg/m2 < body mass index < 37.5 kg/m2; Class 2 obesity: body mass index > 37.5 kg/m2.

CONTACTS AND LOCATIONS:
Overall Officials: Yuntao Nie, M.D., Study Chair — China-Japan Friendship Hospital
Locations (1):
- Yuntao Nie, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes